CLINICAL TRIAL: NCT05334407
Title: Does the Rehabilitation of Masticatory Function and/or Brief Dietary Advice Improve the Diet and Nutrition of Older Subjects With Terminal Dentition or Full Edentulism? A Factorial Randomized Controlled Clinical Trial
Brief Title: Effect of Implant Treatment and/or Dietary Advice on the Nutrition of Edentulous Ageing Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Maurizio Tonetti, Director of Shanghai Perioimplant Innovation Center，Professor of Shanghai Jiao Tong University School of Medicine, chairman of expert Committee of National Clinical Research Center., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: nutrition2021
Record Dates: First submitted 2022-04-05; First posted 2022-04-19 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Edentulous Jaw; Periodontitis
Keywords: nutrition; implant-supported fixed prosthesis; diet intake; healthy ageing; masticatory function
MeSH Terms: conditions — Jaw, Edentulous; Periodontitis | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design (4 month follow up) and longitudinal follow-up to 12 months
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Timing of treatment will be concealed to the therapist and to the examiners. All laboratory assessments will be performed blindly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GroupA（DE+/DI+） (Experimental): The treatment includes the combination of implant-supported full-arch fixed prostheses (dental intervention, DE) and dietary intervention tailored to the dental status (dietary intervention, DI) without waiting period
  Interventions: Procedure: Implant-supported full-arch fixed dental prostheses（dental intervention,DE）; Behavioral: Dietary intervention tailored to the dental status (dietary intervention, DI)
- GroupB（DE+/DI-） (Active Comparator): The treatment includes implant-supported full-arch fixed prostheses (dental intervention, DE) without waiting period and dietary intervention tailored to the dental status (dietary intervention, DI) 4-month later
  Interventions: Procedure: Implant-supported full-arch fixed dental prostheses（dental intervention,DE）; Behavioral: Delayed dietary intervention tailored to the dental status (dietary intervention, DI)
- GroupC（DE-/DI+） (Active Comparator): The treatment includes dietary intervention tailored to the dental status (dietary intervention, DI) without waiting period and implant-supported full-arch fixed prostheses (dental intervention, DE) 4-month later
  Interventions: Behavioral: Dietary intervention tailored to the dental status (dietary intervention, DI); Procedure: Delayed implant-supported full-arch fixed dental prostheses（dental intervention,DE）
- GroupD（DE-/DI-） (Placebo Comparator): The treatment included implant-supported full-arch fixed prostheses (dental intervention, DE) and dietary intervention tailored to the dental status (dietary intervention, DI) with 4-month waiting period. Only general dietary information is provided at baseline.
  Interventions: Procedure: Delayed implant-supported full-arch fixed dental prostheses（dental intervention,DE）; Behavioral: Delayed dietary intervention tailored to the dental status (dietary intervention, DI)

INTERVENTIONS:
Procedure: Implant-supported full-arch fixed dental prostheses（dental intervention,DE） — Implant-supported full-arch fixed dental prostheses in at least one jaw and appropriate treatment in the opposing jaw regarding periodontal diseases, caries, replacement of missing teeth and soft tissue disorders to get at least 10 pairs of occluding teeth. The intervention is designed to provide rehabilitation of masticatory function.
  Other Names: Immediate rehabilitation of masticatory function
  Arms: GroupA（DE+/DI+）; GroupB（DE+/DI-）
Behavioral: Dietary intervention tailored to the dental status (dietary intervention, DI) — Dietary intervention based on the health Belief Model (HBM) with the behavioral goal of increasing an individual's likelihood of food intake regarding fresh vegetables, fresh fruits, and high quality protein for the potential intervention strategies.
  Participants will receive 20 minutes' coordinated dietary advice in the form of the slideshow presentation . A pamphlet prepared with reference to the Supplementary Guidelines for Elderly Populations, the 4th edition of the Dietary Guidelines for Chinese will be given to the participant separately. If a participant does not prepare his or her own meals, the person who does the cooking receives the dietary advice as well.
  Other Names: Immediate dietary intervention
  Arms: GroupA（DE+/DI+）; GroupC（DE-/DI+）
Procedure: Delayed implant-supported full-arch fixed dental prostheses（dental intervention,DE） — Delayed (4 months) implant-supported full-arch fixed dental prostheses in at least one jaw and appropriate treatment in the opposing jaw regarding periodontal diseases, caries, replacement of missing teeth and soft tissue disorders to get at least 10 pairs of occluding teeth. The intervention is designed to provide rehabilitation of masticatory function.
  Other Names: Delayed rehabilitation of masticatory function
  Arms: GroupC（DE-/DI+）; GroupD（DE-/DI-）
Behavioral: Delayed dietary intervention tailored to the dental status (dietary intervention, DI) — Dietary intervention based on the health Belief Model (HBM) with the behavioral goal of increasing an individual's likelihood of food intake regarding fresh vegetables, fresh fruits, and high quality protein for the potential intervention strategies.
  Participants will receive 20 minutes' coordinated dietary advice in the form of the slideshow presentation . A pamphlet prepared with reference to the Supplementary Guidelines for Elderly Populations, the 4th edition of the Dietary Guidelines for Chinese will be given to the participant separately. If a participant does not prepare his or her own meals, the person who does the cooking receives the dietary advice as well.
  Other Names: Delayed dietary intervention
  Arms: GroupB（DE+/DI-）; GroupD（DE-/DI-）

SUMMARY:
Loss of masticatory function consequent to tooth loss is associated with changes in food choices and insufficient nutrition intake. To date, studies showed no significant improvement in nutrient intake with interventions based solely on dental prostheses. Pilot studies have shown positive impacts of interventions combining implant-supported fixed dental prosthesis with brief dietary interventions. The relative contribution and the potential synergy of the components of such interventions need to be determined as it has major public health implications for the community-dwelling ageing population that continues to disproportionately suffer from tooth loss and its consequences.

This study tests the effect of rehabilitation of masticatory function with fixed implant supported dentures and diet re-education on the dietary intake and nutrition in older subjects with terminal dentition (stage IV periodontitis) or full edentulism.

A 2 × 2 factorial randomized controlled trial of eligible adult (≥60 years) with loss of masticatory function consequent to full arch edentulism or terminal dentition (n = 120) will be conducted to test whether the rehabilitation of masticatory function with fixed implant supported dentures, diet re-education and/or their combination improves the diet and nutrition of ageing subjects. The study has been designed to detect changes in fruit and vegetable intake at 4 months using the 24-hour dietary recall method. Changes in protein as percentage of total energy, nutritional biomarkers, metabolomics, oral and gut microbiome, quality of life and masticatory function will also be assessed.

DETAILED DESCRIPTION:
Complete edentulism or presence of a terminal dentition that is functionally compromised in an irreparable way represent the end of the spectrum of caries and periodontitis, eventually leading to loss of masticatory function. These subjects tend to show change in their diet behavior choosing softer diets with higher carbohydrates and fat and less fresh fruit and vegetables.

Accumulating evidence points to the presence of an association between changes in dietary behavior consequent to tooth loss and insufficient nutrition intake. Such impaired nutrition may have long term effects on muscle strength and physical decline, and be detrimental to general health. Indeed, the recent GBD study of dietary risk factors identifies 15 important disease associated exposures. Their analysis shows that 5 of the health associated exposures: consumption of fruit, vegetables, whole grains, nuts, and fiber require a good level of mastication.

While the physiology of mastication is an essential component of alimentation and contributes to the broader process of nutrition, a more holistic approach is needed to properly establish the scientific basis of the contribution of oral health to nutrition and healthy ageing. Assuming a potential cause-effect relationship between the inadequate food choice consequent to tooth loss and compromised nutrition intake, several studies have tried to improve the nutrient intake among edentulous individuals with various types of dentures. However, this goal has not been readily achieved with either complete denture or implant-retained overdenture, given the function limitation on these prosthesis and the lack of dietary intervention.

A small-scale case series has shown that implant-supported fixed prosthesis resulted in more efficient mastication and improved nutrient intake compared with conventional and implant-based removable dentures in partial edentulism. However, no evidence is available regarding the effect of re-establishment of masticatory function with an implant-supported fixed prosthesis in edentulous patients.

Moreover, with the increasing evidence suggesting a positive impact of nutrition counselling on the dietary intake, brief dietary advice has been advocated to help patients make full use of the enhanced masticatory function to improve their diet. Ellis et al. further showed that the impact of dietary advice on patient's satisfaction with dentures and oral health-related quality of life depends on the nature of the prosthesis. No trial has been performed to assess the benefit of dietary advice only or the combined effect of re-establishment of masticatory function with an implant-supported fixed prosthesis and dietary advice in edentulous elderly subjects.

This is a 2 × 2 factorial clinical trial aimed to assess the effect of rehabilitation of masticatory function with fixed implant supported dentures and simultaneous diet re-education on the diet intake and nutrition in ageing subjects with terminal dentition (stage IV periodontitis) or full edentulism.

ELIGIBILITY:
Inclusion Criteria:

* being edentulous or having the presence of terminal dentition (defined as few remaining teeth insufficient in terms of number, position and health status to provide adequate anchorage to a tooth supported or a tooth retained denture) and looking for implant-supported fixed denture treatment
* accepted treatment plan for fixed implant-supported prosthesis restoring at least 10 pairs of occluding teeth
* self-reported inadequate vegetable or fruit or protein intakes (patients were included if at least one of the three criteria listed below were met) I. Patients with a total average daily intake of < 80 g of poultry, meat and aquatic product. II. Patients with an average daily intake of < 200 g of fruit. III. Patients with an average daily intake of < 300 g of vegetables.
* understand written and spoken Chinese and who could respond to Chinese questionnaires
* able and willing to give informed consent for participation in the study
* able and willing to comply with 12-month follow-up

Exclusion Criteria:

* general contraindications to elective oral surgery procedures
* local contraindications to implant-supported immediate-loading fixed prosthesis (e.g. limited jaw opening, insufficient bone volumes/densities)
* looking for replacement of existing implant-retained overdenture with implant-supported fixed denture treatment
* presence of infectious disease, acute or chronic symptoms of TMJ disorder
* psychiatric disorder, dementia
* any dietary restriction, currently taking nutrient supplements or inability to choose his/her diet.
* uncontrolled diabetes (HbA1c≥7.0%)
* self-reported heavy smokers (>10 cigarette/day)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
changes in intake of fruit and vegetables | from baseline to 4-month
  Three 24-hour dietary recall will be conducted through interview, twice on weekdays and once on weekend. The data on food consumption will be converted into the corresponding nutrient contents based on the China Food Composition Tables Standard Edition

SECONDARY OUTCOMES:
Nutrient intake | at baseline, 4, 8, 12 and 16 months
  The intake of fruit and vegetables, protein% of total energy according to a modified version of food-frequency questionnaire
Masticatory function | at baseline, 4, 8, 12 and 16 months
  Ability to mix a two-color chewing gum with 20 masticatory cycles. The obtained bolus will be pressed to a standardized height and a color image will be acquired. Quantitative data will be obtained by digital analysis of the image using variance of hue as the outcome
Peri-implant oral hygiene | at 4, 8, 12 and 16 months for groups with implants
  Modified plaque index (mPI) measured by periodontal probing
Peri-implant soft and hard tissue health (probing depth) | at 4, 8, 12 and 16 months for groups with implants
  Peri-implant probing depth (PD) measured by periodontal probing
Peri-implant soft and hard tissue health (local inflammation) | at 4, 8, 12 and 16 months for groups with implants
  Peri-implant modified bleeding index (mBI) measured by periodontal probing
Peri-implant radiographic bone level stability | 4, and 12 months after dental implant placement (in the context of standard care)
  Standardized panoramic radiographic imaging will be conducted to assess the peri-implant bone level.
OHIP-14 questionnaire | at baseline, 4, 8, 12 and 16 months
  the impact of oral health on the quality of life of participants assessed with the oral health impact profile (OHIP)-14. A 5-point scale was used to calculate the score for each of 14 items. The total score of OHIP-14 is in the range of 0 to 56 with higher values indicating more frequent impacts
Metabolism and systemic inflammatory biomarkers (i) | at baseline, 4, 8, 12 and 16 months
  blood plasma concentration of homocysteine (gas chromatography)
Metabolism and systemic inflammatory biomarkers (ii) | at baseline, 4, 8, 12 and 16 months
  Plasma hs-CRP assessed by immunoturbidometry
Metabolism and systemic inflammatory biomarkers (iii) | at baseline, 4, 8, 12 and 16 months
  Plasma TNF-α (ELISA)
Metabolism and systemic inflammatory biomarkers (iv) | at baseline, 4, 8, 12 and 16 months
  Plasma IL-1β (ELISA)
Metabolism and systemic inflammatory biomarkers (v) | at baseline, 4, 8, 12 and 16 months
  Plasma IL-6 (ELISA)
Oxidative stress biomarkers (i) | at baseline, 4, 8, 12 and 16 months
  Plasma Co Q10 with liquid chromatography-mass spectrometry
Oxidative stress biomarkers (ii) | at baseline, 4, 8, 12 and 16 months
  Plasma uric acid (the enzymatic method)
Oxidative stress biomarkers (iii) | at baseline, 4, 8, 12 and 16 months
  Plasma superoxide dismutase (the chemical colorimetric method)
Nutritional biomarker（Plasma vitamin A） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma vitamin A assessed by liquid chromatography-mass spectrometry
Nutritional biomarker（Plasma vitamin B2） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma vitamin B2 assessed by liquid chromatography-mass spectrometry
Nutritional biomarker（Plasma vitamin B12） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma vitamin B12 assessed by liquid chromatography-mass spectrometry
Nutritional biomarker（Plasma folate） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma folate assessed by liquid chromatography-mass spectrometry
Nutritional biomarker（Plasma vitamin C） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma vitamin C assessed by liquid chromatography-mass spectrometry
Nutritional biomarker（Plasma vitamin E） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma vitamin E assessed by liquid chromatography-mass spectrometry
Nutritional biomarker（plasma α-carotene） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma α-carotene assessed by liquid chromatography-mass spectrometry
Nutritional biomarker（plasma β-carotene） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma α-carotene assessed by liquid chromatography-mass spectrometry
Nutritional biomarker（plasma β-cryptoxanthin） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma β-cryptoxanthin assessed by liquid chromatography-mass spectrometry
Nutritional biomarker（plasma lycopene） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma lycopene assessed by liquid chromatography-mass spectrometry
Nutritional biomarker（plasma lutein/zeaxanthin） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma lutein/zeaxanthin assessed by liquid chromatography-mass spectrometry
Nutritional biomarker（plasma α-tocopherols） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma α-tocopherols assessed by liquid chromatography-mass spectrometry
Nutritional biomarker（plasma γ-tocopherols） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma γ-tocopherols assessed by liquid chromatography-mass spectrometry
Nutritional biomarker（Plasma total cholesterol） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma total cholesterol (Enzymatic Measurements)
Nutritional biomarker（Plasma HDL cholesterol） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma HDL cholesterol (Enzymatic Measurements)
Nutritional biomarker（Plasma LDL cholesterol） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma LDL cholesterol (Enzymatic Measurements)
Nutritional biomarker（Plasma triglycerides） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma triglycerides (Enzymatic Measurements)
Nutritional biomarker（Plasma Lpa） | at baseline, 4, 8, 12 and 16 months
  concentration of plasma Lpa (Enzymatic Measurements)
Metabolomics (Metabolites) | at baseline, 4, 8, 12 and 16 months
  Profiling of annotated plasma metabolites (Differential plasma metabolites with P-value< 0.05 and fold change≥2 or FC≤0.5) based on untargeted metabolomics using liquid chromatography coupled with mass spectrometry analyses
Metabolomics (Oxylipidomics) | at baseline, 4, 8, 12 and 16 months
  Profiling of annotated plasma lipid metabolites (Differential lipid metabolites with P-value< 0.05 and fold change≥2 or FC≤0.5) based on untargeted metabolomics using liquid chromatography coupled with mass spectrometry analyses
Microbiome Analysis(saliva) | at baseline, 4, 8, 12 and 16 months
  Taxonomic profiling with 16S rRNA gene sequencing in saliva samples
Microbiome Analysis(plaque) | at baseline, 4, 8, 12 and 16 months
  Taxonomic profiling with 16S rRNA gene sequencing in subgingival plaque samples
Microbiome Analysis(stool) | at baseline, 4, 8, 12 and 16 months
  Taxonomic profiling with 16S rRNA gene sequencing in stool samples
Nutritional status | at baseline, 4, 8, 12 and 16 months
  assessment by Mini-nutrient status form with a score of 12-14 corresponding to normal nutritional status；8-11 at risk of malnutrition；0-7 malnourished
Muscle strength | at baseline, 4, 8, 12 and 16 months
  muscle strength assessed by Hand grip dynamometer
Cognitive function(i) | at baseline, 4, 8, 12 and 16 months
  cognitive function assessed with the Mini-Mental State Examination with a total score of 30. Score 27-30: normal cognition；Score 21-26: mild cognitive impairment；Score 10-20: moderate cognitive impairment；Score <10: severe cognitive impairment
Cognitive function(ii) | at baseline, 4, 8, 12 and 16 months
  dementia screening with the Alzheimer's disease eight-item tool. With Score 0: no cognitive impairment, Score 1-2: cognitive impairment; Score>=3: dementia
Depression symptoms | at baseline, 4, 8, 12 and 16 months
  assessment with the shortened Center for Epidemiologic Studies Depression Scale. The total score is the sum of 10 items. A score equal to or above 10 is considered depressed.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Tonetti, DMD,PhD, Principal Investigator — Shanghai Perioimplant Innovation Center
Locations (1):
- Shanghai Perio-Implant Innovation Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Result] Kaiser MJ, Bauer JM, Ramsch C, Uter W, Guigoz Y, Cederholm T, Thomas DR, Anthony P, Charlton KE, Maggio M, Tsai AC, Grathwohl D, Vellas B, Sieber CC; MNA-International Group. Validation of the Mini Nutritional Assessment short-form (MNA-SF): a practical tool for identification of nutritional status. J Nutr Health Aging. 2009 Nov;13(9):782-8. doi: 10.1007/s12603-009-0214-7. PMID 19812868
- [Result] Deng K, Uy SNMR, Fok C, Fok MR, Pelekos G, Tonetti MS. Assessment of masticatory function in the differential diagnosis of Stage IV periodontitis: A pilot diagnostic accuracy study. J Periodontol. 2022 Jun;93(6):803-813. doi: 10.1002/JPER.21-0660. Epub 2022 Mar 24. PMID 35239983
- [Result] Ellis JS, Elfeky AF, Moynihan PJ, Seal C, Hyland RM, Thomason M. The impact of dietary advice on edentulous adults' denture satisfaction and oral health-related quality of life 6 months after intervention. Clin Oral Implants Res. 2010 Apr 1;21(4):386-91. doi: 10.1111/j.1600-0501.2009.01859.x. Epub 2010 Jan 22. PMID 20105193
- [Derived] Qian SJ, Liu B, Shi J, Zhang X, Deng K, Shen J, Tao Y, Qiao S, Lai HC, Yuan C, Tonetti MS. Effects of Dental Implants and Nutrition on Elderly Edentulous Subjects: Protocol for a Factorial Randomized Clinical Trial. Front Nutr. 2022 Jun 27;9:930023. doi: 10.3389/fnut.2022.930023. eCollection 2022. PMID 35832045